CLINICAL TRIAL: NCT02145884
Title: Topical Timolol Gel for the Treatment of Infantile Hemangiomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rady Children's Hospital, San Diego (Other)
Collaborators: Valeant Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Sheila Friedlander, MD, Rady Children's Hospital, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PED3560; 20132793 (Other: ICN Pharmaceuticals)
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Hemangioma
Keywords: hemangioma; birthmark; strawberry hemangioma; timolol
MeSH Terms: conditions — Hemangioma; Hemangioma, Cavernous | interventions — Timolol; Gels

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No

ARMS (1):
- timolol maleate 0.5% gel (Experimental): timolol gel 1 to 2 drops twice a day to lesions for 4 months
  Interventions: Drug: timolol maleate 0.5% gel

INTERVENTIONS:
Drug: timolol maleate 0.5% gel — Apply timolol gel 1-2 drops twice a day to lesion
  Other Names: timoptic

SUMMARY:
We plan to conduct a study, to see how safe and effective timolol maleate 0.5% gel-forming solution is for infantile hemangiomas (IH) and the response of hemangiomas to timolol maleate 0.5% . Our hypothesis is that timolol will inhibit and possibly reverse growth of appropriate infantile hemangiomas.

DETAILED DESCRIPTION:
Subjects will be assigned to open label timolol maleate 0.5%. Parents will be instructed to place 1 to 2 drops twice a day in the center of the hemangioma. Subjects are expected to use the study drug as directed every day for a 4 month period.

Subjects will be assessed at baseline, 2 weeks, 4 weeks, and every 4 weeks thereafter for a total of 5 months. Physical exam, photographs to compare size and color intensity, and a scale of improvement will be completed at each visit. Parents will complete a quality of life questionnaire regarding their child's hemangioma and its impact on quality of life.

Subjects who have evidence of worsening would be removed from the study and transferred to the clinic for evaluation and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed permission for study participation and the use of the patient's images are obtained from the patient's parent(s) or guardian(s),

  * The patient is between 7 days and 6 months of age at the time of enrollment,
  * and a proliferating HOI not requiring systemic therapy is present anywhere on the body, Multiple hemangiomas may be treated on same child, if the hemangioma meets this criteria.

Exclusion Criteria:

* patients who are not otherwise generally healthy;
* at risk for imminent ulceration, life-threatening, function-threatening, or ulcerated;
* patients who have previously received systemic, intra-lesional or topical corticosteroids, imiquimod, vincristine, alpha-interferon, propranolol or other beta blockers;
* patients who have previously been treated for his/her HOI, including any surgical and/or medical procedures;
* patients whose mothers have been breastfeeding the patient while also being treated with beta-blockers, systemic corticosteroids, vincristine or alpha-interferon;
* patients who have previously experienced any anaphylactic reactions; patients with an unclear diagnosis of HOI;
* patients participating in another clinical study or living in the same household as an infant already participating in this study;
* patients born prematurely who have not yet reached his/her term equivalent age; and patients with parent(s) or guardian(s) who cannot be contacted by telephone in case of emergency.

Ages: 7 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in size of hemangioma | Baseline, week 2, 4, 8, 12, 16
  At each visit, the size of the IH is assessed in three dimensions (length, width, and height) in cm.
Change in color of hemangioma | Baseline, week 2, 4, 8, 12, 16
  At each visit, the color intensity (e.g., barely perceptible; pale pink or mottled pink/red; red with central pallor; dull red; bright red) of the IH is assessed on a 6 point scale.

SECONDARY OUTCOMES:
Measure the extent of systemic absorption and the factors which influence absorption | week 2
  A heel stick blood sample is collected to assess for systemic absorption.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila F Friedlander, MD, Principal Investigator — Rady Children's Hospital/ University of California, San Diego
Locations (1):
- Pediatric and Adolescent Dermatology, Rady Children's Hospital/University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes